CLINICAL TRIAL: NCT02686060
Title: In-line Filtration to Reduce Systemic Inflammatory Response Syndrome in Babies Born Very prEtErm
Acronym: FRISBEE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2015-A01307-42
Record Dates: First submitted 2016-02-15; First posted 2016-02-19 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2018-02

CONDITIONS: Babies Born Very Preterm

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- in-line filters (Experimental): 0.2 micron positively charged PALL Corporation filters for parenteral nutrition (Posidyne® NEO Intravenous Filter Set) and 1.2 micro IV in-line filters used for lipid administration (Lipipor™ NEO Filters for Neonatal Parenteral Nutrition)
  Interventions: Device: 0.2 micron positively charged PALL Corporation filters and 1.2 micro IV in-line filters used for lipid administration
- without in-line filters. (No Intervention)

INTERVENTIONS:
Device: 0.2 micron positively charged PALL Corporation filters and 1.2 micro IV in-line filters used for lipid administration
  Arms: in-line filters

SUMMARY:
While venous access is an essential part of caring for the preterm neonate potential severe adverse events, including contamination of fluids with bacteria, endotoxins and particulates could occur (Bethune 2001).

Infusion therapy carries a risk for catheter-associated septicaemia (Geiss 1992) originated from the catheter tubing, the ports, at the cannula site or from contaminated infusion fluid. While not all infections lead to septicaemia, immuno-compromised patients such as neonates are at greater risk, and infection becomes a major problem (Ng 1989) and a major risk factor for neurodevelopmental disabilities (Volpe 2008). Indeed, it has been postulated that endotoxins may be involved in the pathogenesis of a proportion of cases of periventricular leukomalacia, the most frequent brain damage associated with neurocognitive handicaps in the human neonate (Volpe 2001).

The presence of calcium in parenteral nutrition mixture leads to precipitation due to its incompatibility with the other components of the admixtures and leads to high concentration of particles (Athanasiou 2014). Adverse systemic effects of particulate matter including phlebitis, granulomata formation in the lung (Marshall 1987) and ischaemic necrosis, are a common finding in necrotizing enterocolitis another serious complication flowing preterm birth (Ballance 1990). Particle contamination of infusion solutions exists despite a stringent infusion regiment. The number and composition of particles depends on the complexity of the applied admixtures (Jack 2010).

Particulate contamination is due to drug incompatibility reactions or their incomplete reconstitution during the preparation process (Schroder 1994). Various studies have demonstrated the contamination of infusion solutions with glass particles from opening glass ampoules, particles from rubber stoppers or conglomerates of the parenteral nutrition components (Ball 2003). Particles have also been shown to be inherent to generic drug formulation (Oie 2005). In an intensive care setting the particle burden may rise up to one million infused particles per day, increasing with the complexity and quantity of the administered infusions (Walpot 1989).

There are two main IV filter pore sizes; the 0.2 micron filter is used for aqueous solutions, and the 1.2 micron filter is recommended for larger molecule solutions such as lipids. The 0.2 micron filter has also been reported to remove air, microorganisms and particulate matter. In addition, endotoxin retention is reportedly achieved by using a positively charged filter membrane; toxic macro-molecules are released by gram-negative bacteria and are claimed to be effective for up to ninety six hours (Bethune 2001).

In-line IV filters are currently claimed to be an effective strategy for the removal of bacteria, endotoxins and particulates associated with intravenous therapy in adults (Ball 2003) and particularly effective in the removal of particles caused from drug precipitate such as antibiotics (Chee 2002; Ball 2003).

However, evidence of the beneficial effect of in-line IV filters in children and neonates is much weaker, despite some positive studies (Jack 2012; Boehne 2013; Sasse 2015). In the population of preterm infants, no study is currently available while particulate contamination due to infusion therapy carries a higher health risk in this subpopulation.

The benefits of using IV in-line filters in critically-ill preterm neonates remains to be demonstrated. This intervention in adults has also been challenged by several authors (Pearson 1996; Newell 1998). Friedland reported that certain drugs such as antibiotics may be retained in the filters causing a reduction in potency (Friedland 1985). On the other hand, there are no known adverse effects from the use of IV in-line filters.

DETAILED DESCRIPTION:
While venous access is an essential part of caring for the preterm neonate potential severe adverse events, including contamination of fluids with bacteria, endotoxins and particulates could occur (Bethune 2001).

Infusion therapy carries a risk for catheter-associated septicaemia (Geiss 1992) originated from the catheter tubing, the ports, at the cannula site or from contaminated infusion fluid. While not all infections lead to septicaemia, immuno-compromised patients such as neonates are at greater risk, and infection becomes a major problem (Ng 1989) and a major risk factor for neurodevelopmental disabilities (Volpe 2008). Indeed, it has been postulated that endotoxins may be involved in the pathogenesis of a proportion of cases of periventricular leukomalacia, the most frequent brain damage associated with neurocognitive handicaps in the human neonate (Volpe 2001).

The presence of calcium in parenteral nutrition mixture leads to precipitation due to its incompatibility with the other components of the admixtures and leads to high concentration of particles (Athanasiou 2014). Adverse systemic effects of particulate matter including phlebitis, granulomata formation in the lung (Marshall 1987) and ischaemic necrosis, are a common finding in necrotizing enterocolitis another serious complication flowing preterm birth (Ballance 1990). Particle contamination of infusion solutions exists despite a stringent infusion regiment. The number and composition of particles depends on the complexity of the applied admixtures (Jack 2010).

Particulate contamination is due to drug incompatibility reactions or their incomplete reconstitution during the preparation process (Schroder 1994). Various studies have demonstrated the contamination of infusion solutions with glass particles from opening glass ampoules, particles from rubber stoppers or conglomerates of the parenteral nutrition components (Ball 2003). Particles have also been shown to be inherent to generic drug formulation (Oie 2005). In an intensive care setting the particle burden may rise up to one million infused particles per day, increasing with the complexity and quantity of the administered infusions (Walpot 1989).

There are two main IV filter pore sizes; the 0.2 micron filter is used for aqueous solutions, and the 1.2 micron filter is recommended for larger molecule solutions such as lipids. The 0.2 micron filter has also been reported to remove air, microorganisms and particulate matter. In addition, endotoxin retention is reportedly achieved by using a positively charged filter membrane; toxic macro-molecules are released by gram-negative bacteria and are claimed to be effective for up to ninety six hours (Bethune 2001).

In-line IV filters are currently claimed to be an effective strategy for the removal of bacteria, endotoxins and particulates associated with intravenous therapy in adults (Ball 2003) and particularly effective in the removal of particles caused from drug precipitate such as antibiotics (Chee 2002; Ball 2003).

However, evidence of the beneficial effect of in-line IV filters in children and neonates is much weaker, despite some positive studies (Jack 2012; Boehne 2013; Sasse 2015). In the population of preterm infants, no study is currently available while particulate contamination due to infusion therapy carries a higher health risk in this subpopulation.

The benefits of using IV in-line filters in critically-ill preterm neonates remains to be demonstrated. This intervention in adults has also been challenged by several authors (Pearson 1996; Newell 1998). Friedland reported that certain drugs such as antibiotics may be retained in the filters causing a reduction in potency (Friedland 1985). On the other hand, there are no known adverse effects from the use of IV in-line filters.

ELIGIBILITY:
Inclusion Criteria:

* Every newborn with a gestational age between 24+0 and 31+6 weeks of gestation or with a birth weight <1500 gm, born at the maternity of Robert Debré children's hospital,
* Neonates whose parental authority holders have been informed for the study & do not opposite to participate,
* Neonates whose parental authority holders are covered by the social security system or CMU.

Exclusion Criteria:

* Preterm infants with a gestational age ≥ 32 weeks of gestation,
* Congenital malformation and/or heart diseases other than patent ductus arteriosus or foramen ovale,
* "Outborn" neonates,
* Newborns whose parental authority holders are minor,
* Newborns with severe birth asphyxia (cord blood pH<7.0 or Apgar score < 5 at 10 min),
* Newborns whose parental authority holders are not beneficiaries of social security coverage.

Ages: 24 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 160 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2017-10-05 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
serum concentrations pattern of 4 major pro-inflammatory cytokines (IL1beta, IL6, IL8 and TNFalpha) | 18 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hopital Robert Debre, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Virlouvet AL, Pansiot J, Toumazi A, Colella M, Capewell A, Guerriero E, Storme T, Rioualen S, Bourmaud A, Biran V, Baud O. In-line filtration in very preterm neonates: a randomized controlled trial. Sci Rep. 2020 Mar 19;10(1):5003. doi: 10.1038/s41598-020-61815-4. PMID 32193413